CLINICAL TRIAL: NCT06209866
Title: The Role Of Global Limb Anatomic Staging System ( GLASS) Compared to Wound, Ischemia, Foot Infection Stage ( WIFI) in Predicting Limb Salvage After Endovascular Revascularization Procedures in Chronic Limb Threatening Ischemia Patients
Brief Title: The Role of Glass Stage Compared to WIFI Stage in Predicting Limb Salvage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Bashandi, Mohamed.15235432@med.aun.edu.eg, Assiut University
Other Study IDs: Glass Stage and WIFI Stage
Record Dates: First submitted 2024-01-06; First posted 2024-01-18 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Chronic Limb-Threatening Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PTA — Percutaneous Trans lumenal Angioplasty

SUMMARY:
compare between GLASS and WIFI Staging in predicting limb salvage in patients with chronic limb threatening ischemia ( CLTI) undergoing endovascular revascularization.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is estimated to affect over 200 million people worldwide. These rates are expected to rise as increasing life expectancies continue to shift the population toward older age. At the most severe end of the disease spectrum, chronic limb-threatening ischemia (CLTI) affects 11% of patients with PAD and is associated with high rates of limb loss and mortality as well as high costs of care.(1) The Society for Vascular Surgery's WIfI (Wound, Ischemia, foot Infection) staging system was developed to classify threatened limbs using factors that affect amputation risk and clinical management in patients with chronic limb threatening ischemia . These include the extent of the wound, degree of ischemia, and severity of any foot infection. It has been validated as a predictor of limb salvage in peripheral artery disease.(2,3)

The Global Vascular guidelines 'GVG "proposes a new Global Anatomic Staging System (GLASS), which is a new method of quantifying the anatomic severity of infrainguinal disease in patients with chronic limb-threatening ischemia. But it has not been used for predicting limb salvage apart from use as a tool in deciding the mode of intervention for patients with chronic limb-threatening ischemia (CLTI).

ELIGIBILITY:
Inclusion Criteria:

-

Patients with CLTI who will undergo endovascular revascularization at our department:

• Rutherford stage 4 ( rest pain) ,stage 5 (ischemic ulceration not exceeding ulcer of the digits of the foot) , stage 6 ( severe ischemic ulcers or frank gangrene)

Exclusion Criteria:

* Rutherford stage 1,2,3 Aortoiliac level of occlusion Unsalvageable limb Patients with contraindications to contrast media Non Atherosclerotic lschemia as • Acute ischemia

  * Post Traumatic Ischemia
  * Chronic ischemia caused by connective tissue diseases or vasculitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at vascular surgery department of Assiut university
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Technical Success | Baseline
  in - line arterial flow to the foot without any flow limiting dissection or residual stenosis > 30% on completion intraoperative arteriography
Time to complete healing | Baseline
  Time to complete healing of the wound after revascularization, Debridement or minor amputation
Limb Salvage | Baseline
  freedom from major amputation above the foot level
Primary Patency | Baseline
  uninterrupted vessel patency with no procedure performed on the treated limb.
Assisted Primary Patency | Baseline
  the percentage of failing but still patent vessel undergoing elective intervention, included patients required revision of the revascularization before vessel occlusion occurs as prophylactic interventions to maintain patency.
Secondary Patency | Baseline
  an occluded artery that required intervention to restore patency.

REFERENCES:
- [Background] Nehler MR, Duval S, Diao L, Annex BH, Hiatt WR, Rogers K, Zakharyan A, Hirsch AT. Epidemiology of peripheral arterial disease and critical limb ischemia in an insured national population. J Vasc Surg. 2014 Sep;60(3):686-95.e2. doi: 10.1016/j.jvs.2014.03.290. Epub 2014 May 10. PMID 24820900
- [Background] Ananthakumar Murugavel, Ajay Savlania, Arunanshu Behera,Mandeep Kang, Comparison of GLASS Stage with WIfI Clinical Staging for Predicting Limb Salvage in Peripheral Arterial Disease.j.jvs.2023.01.104
- [Background] Conte MS, Bradbury AW, Kolh P, White JV, Dick F, Fitridge R, Mills JL, Ricco JB, Suresh KR, Murad MH, Aboyans V, Aksoy M, Alexandrescu VA, Armstrong D, Azuma N, Belch J, Bergoeing M, Bjorck M, Chakfe N, Cheng S, Dawson J, Debus ES, Dueck A, Duval S, Eckstein HH, Ferraresi R, Gambhir R, Gargiulo M, Geraghty P, Goode S, Gray B, Guo W, Gupta PC, Hinchliffe R, Jetty P, Komori K, Lavery L, Liang W, Lookstein R, Menard M, Misra S, Miyata T, Moneta G, Munoa Prado JA, Munoz A, Paolini JE, Patel M, Pomposelli F, Powell R, Robless P, Rogers L, Schanzer A, Schneider P, Taylor S, De Ceniga MV, Veller M, Vermassen F, Wang J, Wang S; GVG Writing Group for the Joint Guidelines of the Society for Vascular Surgery (SVS), European Society for Vascular Surgery (ESVS), and World Federation of Vascular Societies (WFVS). Global Vascular Guidelines on the Management of Chronic Limb-Threatening Ischemia. Eur J Vasc Endovasc Surg. 2019 Jul;58(1S):S1-S109.e33. doi: 10.1016/j.ejvs.2019.05.006. Epub 2019 Jun 8. PMID 31182334
- [Background] Mills JL Sr, Conte MS, Armstrong DG, Pomposelli FB, Schanzer A, Sidawy AN, Andros G; Society for Vascular Surgery Lower Extremity Guidelines Committee. The Society for Vascular Surgery Lower Extremity Threatened Limb Classification System: risk stratification based on wound, ischemia, and foot infection (WIfI). J Vasc Surg. 2014 Jan;59(1):220-34.e1-2. doi: 10.1016/j.jvs.2013.08.003. Epub 2013 Oct 12. PMID 24126108